CLINICAL TRIAL: NCT04694053
Title: Fournier's Gangrene as a Rare Complication in Patient With Uncontrolled Type 2 Diabetes Treated With Surgical Debridement: a Case Report and Literature Review
Brief Title: Fournier's Gangrene in Patient With Uncontrolled Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Daniele Provenzano, Principal Investigator, University of Catania
Other Study IDs: Clinica Ch 1
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Fournier Gangrene
Keywords: Fournier's gangrene; Type 2 diabetes; surgical debridement
MeSH Terms: conditions — Fournier Gangrene; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical debridement — The surgical team performed an extended surgical debridement to healthy tissue of external genital, as well as perineal, perianal, and infrapubic regions.

SUMMARY:
A 66-year-old man, with a history of uncontrolled type 2 diabetes, obesity with BMI 38, chronic kidney failure and chronic heart failure, was admitted to the Emergency Department with a large area of necrosis involving the perineal and perianal regions.

DETAILED DESCRIPTION:
Fournier's gangrene is a potentially fatal emergency condition, supported by an infection of perineal and perianal region, characterized by necrotizing fasciitis with a rapid spread to fascial planes. FG, usually due to compromised host, may be sustained by many microbial pathogens.

A 66-year-old man, with a history of uncontrolled type 2 diabetes, obesity with BMI 38, chronic kidney failure and chronic heart failure, was admitted to the Emergency Department with a large area of necrosis involving the perineal and perianal regions.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Fournier's Gangrene Insulin dependent diabetes (type 2)

Exclusion Criteria:

n/a

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A 66-year-old man, with a history of uncontrolled type 2 diabetes, obesity with BMI 38, chronic kidney failure and chronic heart failure, was admitted to the Emergency Department with a large area of necrosis involving the perineal and perianal regions.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants | From 3 November 2020 at 23 November 2020
  Number of patients enrolled by the emergency room.
Fournier's gangrene evolution after treatment | 20 days
  Evolution of gangrene after surgical debridement of perineal and perianal regions.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele o Provenzano, md, Principal Investigator — https://www.unict.it/
Locations (1):
- University of Catania, Catania, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT04694053/Prot_000.pdf